CLINICAL TRIAL: NCT01656512
Title: Analysis of Outcome of Bisphosphonate Use in Children With ALL- "Case Controlled Study"
Brief Title: Zometa Study in Pediatric Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Cancer Hospital Egypt 57357 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCHE-ALL002
Record Dates: First submitted 2012-07-30; First posted 2012-08-03 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Osteoporosis
Keywords: ALL; zoledronic acid; Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Diphosphonates; Calcium; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm ( A) (Active Comparator): Arm ( A) : patients will receive calcium & vitamin D
  Interventions: Drug: calcium & vitamin D
- Arm (B) (Experimental): we will give calcium and Vitamin D daily in addition to bisphosphonates (zolendronic acid ) every 3 months in the dose of
  Interventions: Drug: zolendronic acid

INTERVENTIONS:
Drug: zolendronic acid — patients will receive calcium & vitamin D daily in addition to bisphosphonates (zolendronic acid ) every 3 months in the dose of
  1. Initial dose: (0.025) mg /kg
  2. Subsequent doses ( 0.05) mg /kg.
  3. Maximum dose of 4 mg.
  Other Names: bisphosphonates
  Arms: Arm (B)
Drug: calcium & vitamin D — patients will receive calcium & vitamin D Dose of Calcium : 1500- 2000 gram elemental Calcium daily . Dose of Vitamin D ( calcitriol; one alpha) 800-1000 International Unit
  Arms: Arm ( A)

SUMMARY:
Acute Lymphoblastic Leukemia (ALL) is the most common malignancy in children. It accounts for one fourth of all childhood cancers & 74 % of childhood leukemia. Based upon drug registry data, children prescribed more than three courses of systemic glucocorticoids yearly faced a 20% increase in age-adjusted fracture rates. Rapid recovery occurred once glucocorticoids were discontinued, and fracture rates returned to expected for age by 1 year after treatment (Journal Of Clinical Endocrinology & Metabolism 2009). The investigators will study the role of bisphosphonates in the prevention of secondary osteoporosis in children & adolescents treated for ALL in the Children's Cancer Hospital -Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Age above 5 & below 18 years at the time of diagnosis.
* Newly diagnosed ALL patients.
* Not previously treated, previous steroid intake not more than 72 hours.
* Treated according to St Judy study XV protocol.

Exclusion Criteria:

* Previous steroid intake more than 72 hours.
* Less than 5 years

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 95 (Actual)
Dates: Start 2011-10; Primary Completion 2014-01 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Measure the change in the Bone densitometry due to secondary osteoporosis | 1- At baseline ( not more than 48 hours of start of therapy with steroids) 2- At week 48 3- At end of treatment ( week 120 for girls ) & ( week 146 for boys) 4-As required clinically eg: fractures .
  we will do the following for evaluation :
  1. Bone densitometry using Dual-energy x-ray absorptiometry (DXA) scan analyzed using the Z-score. To be done :
     * At baseline ( not more than 48 hours of start of therapy with steroids)
     * At week 48
     * At end of treatment ( week 120 for girls ) & ( week 146 for boys)
     * As required clinically eg: fractures .
  2. Magnetic resonance imaging of both hips & knees will be done at reinduction I & II & if symptomatic.

SECONDARY OUTCOMES:
- To assess the percentage change in lumbar spine BMD at wk 48 relative to baseline in both arms. | week 48 continuation phase

CONTACTS AND LOCATIONS:
Overall Officials: Shimaa Samir, MBBCH, Principal Investigator — Children's Cancer Hospital Egypt 57357
Locations (1):
- Children's Cancer Hospital Egypt 57357, Cairo, Egypt